CLINICAL TRIAL: NCT05636436
Title: A Phase I, Single Center, Randomized, Blinded, Controlled Clinical Trial to Evaluate the Safety, Tolerability and Preliminary Immunogenicity of Recombinant Herpes Zoster Vaccine (CHO Cells) in Healthy Subjects Aged 18 Years and Above
Brief Title: Safety and Immunogenicity of Recombinant Herpes Zoster Vaccine (CHO Cells) in Healthy Subjects Aged 18 Years and Above
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: MAXVAX Biotechnology Limited Liability Company (Industry)
Collaborators: Henan Center for Disease Control and Prevention (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: MKKCT-100-001
Record Dates: First submitted 2022-11-16; First posted 2022-12-05 (Actual); Last update posted 2024-11-20 (Actual); Status verified 2024-11

CONDITIONS: Herpes Zoster
MeSH Terms: conditions — Herpes Zoster | interventions — Adjuvants, Pharmaceutic; Sodium Chloride; Injections

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (11):
- Low dose vaccine group in adults aged 18 to 49 years (Experimental): Subjects aged 18 to 49 years will be vaccinated with 2 doses of low dose recombinant herpes zoster vaccine (CHO cells) on a 0, 2 month schedule, administered intramuscularly (IM).
  Interventions: Biological: Low Dose Recombinant Herpes Zoster Vaccine (CHO cells)
- Low dose adjuvant group in adults aged 18 to 49 years (Experimental): Subjects aged 18 to 49 years will be vaccinated with 2 doses of low dose adjuvant on a 0, 2 month schedule, administered intramuscularly (IM).
  Interventions: Biological: Low dose adjuvant
- High dose vaccine group in adults aged 18 to 49 years (Experimental): Subjects aged 18 to 49 years will be vaccinated with 2 doses of high dose recombinant herpes zoster vaccine (CHO cells) on a 0, 2 month schedule, administered intramuscularly (IM).
  Interventions: Biological: High Dose Recombinant Herpes Zoster Vaccine (CHO cells)
- High dose adjuvant group in adults aged 18 to 49 years (Experimental): Subjects aged 18 to 49 years will be vaccinated with 2 doses of high dose adjuvant on a 0, 2 month schedule, administered intramuscularly (IM).
  Interventions: Biological: High dose adjuvant
- Placebo group in adults aged 18 to 49 years (Placebo Comparator): Subjects aged 18 to 49 years will be vaccinated with 2 doses of placebo on a 0, 2 month schedule, administered intramuscularly (IM).
  Interventions: Biological: Placebo
- Low dose vaccine group in adults aged 50 years and older (Experimental): Subjects aged 50 years and older will be vaccinated with 2 doses of low dose recombinant herpes zoster vaccine (CHO cells) on a 0, 2 month schedule, administered intramuscularly (IM).
  Interventions: Biological: Low Dose Recombinant Herpes Zoster Vaccine (CHO cells)
- Low dose adjuvant group in adults aged 50 years and older (Experimental): Subjects aged 50 years and older will be vaccinated with 2 doses of low dose adjuvant on a 0, 2 month schedule, administered intramuscularly (IM).
  Interventions: Biological: Low dose adjuvant
- High dose vaccine group in adults aged 50 years and older (Experimental): Subjects aged 50 years and older will be vaccinated with 2 doses of high dose recombinant herpes zoster vaccine (CHO cells) on a 0, 2 month schedule, administered intramuscularly (IM).
  Interventions: Biological: High Dose Recombinant Herpes Zoster Vaccine (CHO cells)
- High dose adjuvant group in adults aged 50 years and older (Experimental): Subjects aged 50 years and older will be vaccinated with 2 doses of high dose adjuvant on a 0, 2 month schedule, administered intramuscularly (IM).
  Interventions: Biological: High dose adjuvant
- Shingrix® group in adults aged 50 years and older (Active Comparator): Subjects aged 50 years and older will be vaccinated with 2 doses of Shingrix® on a 0, 2 month schedule, administered intramuscularly (IM).
  Interventions: Biological: Positive control
- Placebo group in adults aged 50 years and older (Placebo Comparator): Subjects aged 50 years and older will be vaccinated with 2 doses of placebo on a 0, 2 month schedule, administered intramuscularly (IM).
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: Low Dose Recombinant Herpes Zoster Vaccine (CHO cells) — 0.5 mL per dose, containing a total of 50 µg recombinant varicella zoster virus glycoprotein E, adjuvanted with low dose MA105.
  Arms: Low dose vaccine group in adults aged 18 to 49 years; Low dose vaccine group in adults aged 50 years and older
Biological: High Dose Recombinant Herpes Zoster Vaccine (CHO cells) — 0.5 mL per dose, containing a total of 50 µg recombinant varicella zoster virus glycoprotein E, adjuvanted with high dose MA105.
  Arms: High dose vaccine group in adults aged 18 to 49 years; High dose vaccine group in adults aged 50 years and older
Biological: Low dose adjuvant — 0.5 mL per dose, containing low dose MA105 adjuvant.
  Arms: Low dose adjuvant group in adults aged 18 to 49 years; Low dose adjuvant group in adults aged 50 years and older
Biological: High dose adjuvant — 0.5 mL per dose, containing high dose MA105 adjuvant.
  Arms: High dose adjuvant group in adults aged 18 to 49 years; High dose adjuvant group in adults aged 50 years and older
Biological: Positive control — 0.5 mL per dose, containing a total of 50 µg recombinant varicella zoster virus glycoprotein E, adjuvanted with AS01B.
  Other Names: Shingrix®
  Arms: Shingrix® group in adults aged 50 years and older
Biological: Placebo — 0.5 mL per dose, containing 4.5 mg sodium chloride.
  Other Names: Saline for injection
  Arms: Placebo group in adults aged 18 to 49 years; Placebo group in adults aged 50 years and older

SUMMARY:
The purposes of the study are to evaluate the safety and tolerability of different dose levels of recombinant herpes zoster vaccine (CHO Cells) with 2 doses at 2-month intervals in healthy subjects aged 18 years and older, and to preliminarily explore immunogenicity.

DETAILED DESCRIPTION:
The clinical trial will be a single-center, randomized, blind, controlled study in which two dose levels of vaccine will be tested in healthy adults aged 18 to 49 years and 50 years and older, with progression from low dose level to high dose level and younger age group to the older age group based on assessment of safety and tolerability. The younger cohort (aged 18 to 49 years) will consist of 60 subjects, 30 per dose level, and these 30 subjects will be randomized into three subgroups, including vaccine group, adjuvant group and normal saline group, with randomization ratio of 2:2:1. The older cohort (aged 50 years and older) will consist of 72 subjects, 36 per dose level, and these 36 subjects will be randomized into four subgroups, including vaccine group, adjuvant group, Shingrix® group and normal saline group, with randomization ratio of 2:2:1:1.

ELIGIBILITY:
Inclusion Criteria:

1. Permanent residents aged 18 years and above;
2. Subjects voluntarily agree to participate in the study and signed an informed consent;
3. Be able to participate in all scheduled visits and comply with the protocol requirements.

Exclusion Criteria:

1. Axillary temperature>37.0℃;
2. History of herpes zoster within 5 years before vaccination;
3. Prior vaccination with chickenpox vaccine or herpes zoster vaccine;
4. Female participant who is pregnant ( urine pregnancy test was positive) or breastfeeding, or has pregnancy plans within 1 year after the last vaccination;
5. Receipt of live vaccine within 28 days, or any other vaccine within 14 days prior to vaccination;
6. Receipt of immunoglobulin or intravenous immunoglobulin within 3 months before vaccination;
7. Acute diseases or acute exacerbation of chronic disease within 3 days before vaccination;
8. A known allergy to any components of the study vaccine (especially allergic to aminoglycoside antibiotics), or history of severe allergy to any previous vaccination;
9. History of convulsions, epilepsy, encephalopathy (such as congenital brain dysplasia, brain trauma, brain tumor, cerebral hemorrhage, cerebral infarction, brain infection disease, nerve tissue damage caused by chemical drug poisoning, etc.) or mental illness and family history;
10. Asplenia or functional asplenia, or splenectomy caused by any condition;
11. Primary or secondary impairment of immune function or diagnosed congenital or acquired immunodeficiency, human immunodeficiency virus (HIV) infection, lymphoma, leukemia, systemic lupus erythematosus (SLE), rheumatoid arthritis, juvenile rheumatoid arthritis (JRA), inflammatory bowel disease or other autoimmune diseases;
12. Receipt of immunosuppressive therapy within 3 months before vaccination (such as long-term use of systemic glucocorticoid ≥14 days, dose ≥2mg/kg/day or ≥20mg/day prednisone or equivalent dose), but inhaled, intra-articular and topical steroids are acceptable;
13. Severe cardiovascular disease(eg. Pulmonary heart disease, Pulmonary Edema); Severe liver or kidney disease; or diabetes with complication;
14. History of thrombocytopenia or other coagulation disorders, which may cause intramuscular injection contraindications;
15. Abnormal blood pressure during physical examination before vaccination (systolic pressure ≥ 140 mmHg and/or diastolic pressure ≥ 90 mmHg);
16. Abnormal and clinically significant laboratory test results as determined by the investigator before vaccination;
17. Current or history of alcohol and/or drug abuse;
18. Any condition that, in the opinion the investigator, may affect the safety of the subject or the evaluation of the study results.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 132 (Actual)
Dates: Start 2022-12-07 (Actual); Primary Completion 2024-12-30 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
The incidence and severity of adverse events | Within 30 minutes after each vaccination.
  Incidence and severity of adverse events within 30 minutes after each vaccination. The severity of solicited and unsolicited adverse events will be graded from grade 1 to grade 4, other adverse events will be graded from grade 1 to grade 5.
The incidence and severity of adverse events | Within 7 days after each vaccination.
  Incidence and severity of adverse events within 7 days after each vaccination. The severity of solicited and unsolicited adverse events will be graded from grade 1 to grade 4, other adverse events will be graded from grade 1 to grade 5.
The incidence and severity of adverse events | Day 8 to 30 after each vaccination.
  Incidence and severity of adverse events during Day 8 to 30 after each vaccination. The severity of solicited and unsolicited adverse events will be graded from grade 1 to grade 4, other adverse events will be graded from grade 1 to grade 5.
The incidence and severity of adverse events | Within 30 days after each vaccination.
  Incidence and severity of adverse events within 30 days after each vaccination. The severity of solicited and unsolicited adverse events will be graded from grade 1 to grade 4, other adverse events will be graded from grade 1 to grade 5.
Incidence of abnormal and clinically significant laboratory test results | Day 4 after each vaccination .
  Laboratory test includes hematology, blood biochemistry and urine analysis.

SECONDARY OUTCOMES:
Incidence of Serious Adverse Event | From the first vaccination to 12 months after full vaccination (From Day 0 to Day 420).
  Incidence of Serious Adverse Event (SAE) from the first vaccination to 12 months after full vaccination.
Potential Immune Mediated Disorder | From the first vaccination to 12 months after full vaccination (From Day 0 to Day 420).
  Incidence of Potential Immune Mediated Disorder (pIMD) from the first vaccination to 12 months after full vaccination.
Geometric mean concentration (GMC) of anti-gE antibody and anti-VZV antibody | Prior to each vaccination (Day 0, Day 60).
  Measured by ELISA.
Geometric mean concentration (GMC) of anti-gE antibody and anti-VZV antibody | Day 14 after each vaccination (Day 14, Day 74).
  Measured by ELISA.
Geometric mean concentration (GMC) of anti-gE antibody and anti-VZV antibody | Month 1 after each vaccination (Day 30, Day 90).
  Measured by ELISA.
Geometric mean concentration (GMC) of anti-gE antibody and anti-VZV antibody | Month 6 and 12 after the second vaccination (Day 240, Day 420).
  Measured by ELISA.
Seroconversion rate of anti-gE antibody and anti-VZV antibody | Prior to the second vaccination (Day 60).
  Seroconversion is defined as a ≥4 fold rise in antibody concentration compared with baseline for those antibody concentration was ≥Cut-off value at baseline; or a ≥4 fold Cut-off value in antibody concentration compared with baseline for those antibody concentration was <Cut-off value at baseline.
Seroconversion rate of anti-gE antibody and anti-VZV antibody | Day 14 after each vaccination (Day 14, Day 74).
  Seroconversion is defined as a ≥4 fold rise in antibody concentration compared with baseline for those antibody concentration was ≥Cut-off value at baseline; or a ≥4 fold Cut-off value in antibody concentration compared with baseline for those antibody concentration was <Cut-off value at baseline.
Seroconversion rate of anti-gE antibody and anti-VZV antibody | Month 1 after each vaccination (Day 30, Day 90).
  Seroconversion is defined as a ≥4 fold rise in antibody concentration compared with baseline for those antibody concentration was ≥Cut-off value at baseline; or a ≥4 fold Cut-off value in antibody concentration compared with baseline for those antibody concentration was <Cut-off value at baseline.
Positive rate of anti-gE antibody and anti-VZV antibody | Prior to each vaccination (Day 0, Day 60).
  Positive rate is defined as percentage of subjects with antibody concentration ≥Cut-off value.
Positive rate of anti-gE antibody and anti-VZV antibody | Day 14 after each vaccination (Day 14, Day 74).
  Positive rate is defined as percentage of subjects with antibody concentration ≥Cut-off value.
Positive rate of anti-gE antibody and anti-VZV antibody | Month 1 after each vaccination (Day 30, Day 90).
  Positive rate is defined as percentage of subjects with antibody concentration ≥Cut-off value.
Positive rate of anti-gE antibody and anti-VZV antibody | Month 6 and 12 after the second vaccination (Day 240, Day 420).
  Positive rate is defined as percentage of subjects with antibody concentration ≥Cut-off value.
Geometric mean increase(GMI) of anti-gE antibody and anti-VZV antibody concentration | Prior to the second vaccination (Day 60).
  The antibody concentration prior to the second vaccination compared with that at baseline (Day 0).
Geometric mean increase(GMI) of anti-gE antibody and anti-VZV antibody concentration | Day 14 after each vaccination (Day 14, Day 74).
  The antibody concentration at Day 14 after each vaccination compared with that at baseline (Day 0).
Geometric mean increase(GMI) of anti-gE antibody and anti-VZV antibody concentration | Month 1 after each vaccination (Day 30, Day 90)
  The antibody concentration at 1 month after each vaccination compared with that at baseline (Day 0).
Four-fold increase rate of the anti-gE antibody and anti-VZV antibody concentration | Prior to the second vaccination (Day 60).
  The antibody concentration prior to the second vaccination compared with that at baseline (Day 0).
Four-fold increase rate of the anti-gE antibody and anti-VZV antibody concentration | Day 14 after each vaccination (Day 14, Day 74).
  The antibody concentration at Day 14 after each vaccination compared with that at baseline (Day 0).
Four-fold increase rate of the anti-gE antibody and anti-VZV antibody concentration | Month 1 after each vaccination (Day 30, Day 90).
  The antibody concentration at month 1 after each vaccination compared with that at baseline (Day 0).
Frequency of gE-specific CD4+ T-cells expressing at least 1 Immunological activation marker | Prior to the first vaccination (Day 0).
  The analysis focused on CD4+ T-cells expressing at least 1 immunological activation marker among Interferon gamma (IFN-γ), Interleukin 2 (IL-2), Tumour Necrosis Factor alpha (TNF-α) and CD40 Ligand (CD40L).
Frequency of gE-specific CD4+ T-cells expressing at least 1 Immunological activation marker | Month 1 after the second vaccination (Day 90).
  The analysis focused on CD4+ T-cells expressing at least 1 immunological activation marker among Interferon gamma (IFN-γ), Interleukin 2 (IL-2), Tumour Necrosis Factor alpha (TNF-α) and CD40 Ligand (CD40L).
Frequency of gE-specific CD4+ T-cells expressing at least 1 Immunological activation marker | Month 6, 12 after the second vaccination (Day 240, Day 420).
  The analysis focused on CD4+ T-cells expressing at least 1 immunological activation marker among Interferon gamma (IFN-γ), Interleukin 2 (IL-2), Tumour Necrosis Factor alpha (TNF-α) and CD40 Ligand (CD40L).
Cellular immune response | Prior to the first vaccination (Day 0).
  Cellular immune response is defined as the frequency of gE-specific CD4+ T-cells (expressing at least 1 Immunological activation marker) ≥2 fold increase compared with baseline for those the frequency of gE-specific CD4+ T-cells ≥Cut-off value at baseline; or the frequency of gE-specific CD4+ T-cells (expressing at least 1 Immunological activation marker) ≥Cut-off value for those the frequency of gE-specific CD4+ T-cells <Cut-off value at baseline.
Cellular immune response | Month 1 after the second vaccination (Day 90).
  Cellular immune response is defined as the frequency of gE-specific CD4+ T-cells (expressing at least 1 Immunological activation marker) ≥2 fold increase compared with baseline for those the frequency of gE-specific CD4+ T-cells ≥Cut-off value at baseline; or the frequency of gE-specific CD4+ T-cells (expressing at least 1 Immunological activation marker) ≥Cut-off value for those the frequency of gE-specific CD4+ T-cells <Cut-off value at baseline.
Cellular immune response | Month 6, 12 after the second vaccination (Day 240, Day 420)
  Cellular immune response is defined as the frequency of gE-specific CD4+ T-cells (expressing at least 1 Immunological activation marker) ≥2 fold increase compared with baseline for those the frequency of gE-specific CD4+ T-cells ≥Cut-off value at baseline; or the frequency of gE-specific CD4+ T-cells (expressing at least 1 Immunological activation marker) ≥Cut-off value for those the frequency of gE-specific CD4+ T-cells <Cut-off value at baseline.

CONTACTS AND LOCATIONS:
Overall Officials: Yanxia Wang, Principal Investigator — Henan Center for Disease Control and Prevention
Locations (1):
- Yanjin District Center for Disease Control and Prevention, Xinxiang, Henan, China

IPD SHARING:
Plan to Share IPD: No